CLINICAL TRIAL: NCT05237336
Title: Integrating Psychology of the Soul With Mindfulness-Based Cognitive Therapy for Singapore's Malay Muslims With Psychological Distress: A Mixed-Method Study for Effectiveness and Experience
Brief Title: Integrated Mindfulness-Based Cognitive Therapy for Singapore Malay Muslims
Acronym: IPS-MBCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Islamic University Malaysia (Other)
Responsible Party: Principal Investigator, Jamilah Hanum Abdul Khaiyom, PhD, Assistant Professor, International Islamic University Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IREC 2021-279
Record Dates: First submitted 2022-01-11; First posted 2022-02-14 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Psychological Distress
Keywords: MBCT; Culture; RCT; Islamic
MeSH Terms: interventions — Mindfulness-Based Cognitive Therapy; Counseling

STUDY DESIGN:
Intervention Model Description: This three-group randomised controlled trial recruited 80 Malay Muslims with psychological distress. Participants will be randomly allocated to an MBCT-IPS experimental group, an MBCT group, or individual counselling-as-usual.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MBCT-IPS (Experimental): Mindfulness-based Cognitive Therapy (MBCT) integrated with cultural Psychology of Soul (IPS) 2-session (IPS) + standard 8-session (MBCT)
  Interventions: Behavioral: Mindfulness-based Cognitive Therapy
- Mindfulness-based Cognitive Therapy (Active Comparator): Standard 8-session Mindfulness-based Cognitive Therapy (MBCT)
  Interventions: Behavioral: Mindfulness-based Cognitive Therapy
- Counselling as usual (Other): 8-session Control group
  Interventions: Behavioral: Counselling as usual

INTERVENTIONS:
Behavioral: Mindfulness-based Cognitive Therapy — MBCT is a relapse prevention program that is used to teach participants with chronic physical/mental ailment (used to their conditions):
  * to manage early signs of distresses with compassionate awareness, and respond more effectively to mood and cognitive changes.
  * To become aware of bodily sensations, feelings, and thoughts, from moment to moment.
  * To help participants learn different ways of relating to sensations, thoughts and feelings- through mindful acceptance and acknowledgement of unwanted feelings and thoughts, rather than habitual, automatic, preprogrammed routines that tend to perpetuate difficulties.
  * To help participants to be able to choose the most skilful response to any unpleasant thoughts, feelings or situations that they meet.
  UK's NICE recommends MBCT for persons who are well and have had 3 or more episodes of depression. MBCT benefits persons whose distress is triggered by the way they process experiences.
  Arms: MBCT-IPS; Mindfulness-based Cognitive Therapy
Behavioral: Counselling as usual — Control group, Counselling as usual
  Arms: Counselling as usual

SUMMARY:
Singapore's Institute of Mental Health (IMH) identified the need for culture-based research and clinical intervention catering to the minority populations in Singapore to foster treatment sustainability and recovery. Singapore's Malay population, account for 13.5% of the population. Malays tend to delay or drop-out of psychological treatments that do not address the cultural concerns which they associate to mental illness, i.e., a spiritual disorder caused by character flaws, evil spirits, or religious negligence.

The study examines the effectiveness of Mindfulness-Based Cognitive Therapy - Integrated with Psychology of Soul (MBCT-IPS) with Singaporean Malay Muslims with psychological distress. The secondary aims are to explore their experiences and perceptions on the intervention acceptability, appropriateness, and feasibility. It may provide mental health practitioners with a treatment option that may be integrated with standard therapies.

Methods: This mixed-method, three-group randomised controlled trial recruited 80Malay Muslims with psychological distress at a psychiatric rehabilitation organisation. Participants will be randomly allocated to an MBCT-IPS experimental group, an MBCT group, or individual counselling-as-usual. MBCT-IPS is a 2+8-week group intervention that integrates the Psychology of Soul (IPS) with the standard Mindfulness-Based Cognitive Therapy (MBCT).

General Linear Model (GLM) with an intention-to-treat analysis and per-protocol approach will analyse the study. Participants' and treatment providers' qualitative experiences will be thematically analysed for the acceptability of treatment after the study.

Expected results: Overall improvements in outcome measures are expected with significant differences between groups. Qualitative experiences are hoped to be enriching and therapeutic for both participants and treatment providers, with treatment being appropriate, acceptable, and feasible.

DETAILED DESCRIPTION:
This study examines the effects of MBCT-Integrated with Psychology of Self (IPS), MBCT, and one-on-one counselling-as-usual to reduce symptoms of psychological distress, and increase positive mental health and self-compassion. The IPS combines two modules from the Islamic Religious Council of Singapore (MUIS)'s Adult Islamic Learning (ADIL) programs, the 'An Introduction to Maqasid Syariah' and 'Grief and Suffering', with Dr Abdallah Rothman's grounded theory in Islamic Psychology. The IPS sessions will include Islamic psychoeducation and exercises on purpose, acceptance, letting go, and Islamic concepts on biopsychosocial-spiritual care.

The study also examines whether the participants would consider the intervention appropriate, acceptable, and feasible. We are also interested in exploring participants' understanding and meaning of the intervention and factors contributing to intervention compliance.

Procedure:

Researchers will invite Malay Muslim adults working in the private community, social service organisations, mosques, societies, support groups or studying in higher institutions of learning/universities to participate in the study. They may also invite family and friends to take part in the research. However, participants will not be informed of the various therapies provided or whether their allocation is to the experimental or control groups.

Individuals interested in participating in this study will submit a request online on Qualtrics for researchers to contact them. The Qualtrics form will include the pre-assessment measure Depression, Anxiety, and Stress Scale (DASS-21).

To screen the participants, the researchers will interview potential participants individually online. The interview will (a) assess the participants' suitability utilising the screening questionnaire that includes items for exclusion criteria, (b) readiness for intervention, (c) and informs participants about the process and demands of the study. Informed consent approved by the Agency for Integrated Care (AIC) Institutional Review Board (IRB) will be verbally obtained during the interview. Participants who agree to commit to all the assessment sessions and consent to sessions be recorded will receive the registration link. The online registration form includes a consent form, the participant's demographic information, the 19-item Positive Mental Health (PMH-19), and 12-item Self-Compassion Scale-Short Form (SCS-SF).

Assessments will be conducted on Qualtrics at five points: pre-intervention, fourth week, last session, and follow-up at 1-month & 3-months.

Those who meet the exclusion criteria and are unsuitable for MBCT will be referred to other programs at Club HEAL. Participants may withdraw from intervention at any point before or during intervention and will be contacted for their feedback. Participants who complete the assessments receive honorariums. All participants will be offered the most effective intervention at the end of the study.

Randomisation:

When participants submit their online registration, they will be randomly assigned to an intervention arm. Participants will receive their assignment and schedule via the Qualtrics email distribution.

ELIGIBILITY:
Inclusion Criteria:

1. Must be Malay Muslim, identifying with the Malay race,
2. can speak and understand English,
3. scoring Global Assessment of Functioning (GAF > 61)
4. scoring Mild to Extremely Severe in DASS-21, for at least one subscale of Depression: 5-21; Anxiety: 4-21; Or Stress: 8-21

Exclusion Criteria: Patients (whether inpatient or outpatient) or individuals who report having:

1. a diagnosed mental disorder (schizophrenia, bipolar disorder, & post-traumatic stress disorder or any other mental disorders )
2. psychotic symptoms
3. actively suicidal.
4. personality disorder, including substance use and addiction.
5. neurocognitive disorders or cognitive impairment.
6. persons who have previously undergone structured MBCT treatment or concurrently receiving psychological treatment elsewhere.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Depression, Anxiety, Stress Score (DASS-21) at Week 0 | Week 0
  DASS-21 has twenty-one questions, and is a self-administered survey, measuring core symptoms associated with depression, anxiety, and stress on a four-point Likert scale to indicate each symptom's frequency and intensity for the past week. Ratings begin at 0 as "Never" to 3 for "Almost Always". Depression is interpreted as "normal" when the score is between 0-4, mild at 5-6, moderate at 7-10, severe at 11-13 and extremely severe at 14+. Anxiety is categorised as normal between 0-3, mild at 4-5, moderate at 6-7, severe at 8-9 and extremely severe at 10 or more. Stress is indicated as "normal" between 0-7, "mild" at 8-9, "moderate" at 10-12, severe at 13-16 and extremely severe at 17 or more
Change from Baseline to Depression, Anxiety, Stress Score (DASS-21) at Week 4 | Week 0 and Week 4
  DASS-21 has twenty-one questions, and is a self-administered survey, measuring core symptoms associated with depression, anxiety, and stress on a four-point Likert scale to indicate each symptom's frequency and intensity for the past week. Ratings begin at 0 as "Never" to 3 for "Almost Always". Depression is interpreted as "normal" when the score is between 0-4, mild at 5-6, moderate at 7-10, severe at 11-13 and extremely severe at 14+. Anxiety is categorised as normal between 0-3, mild at 4-5, moderate at 6-7, severe at 8-9 and extremely severe at 10 or more. Stress is indicated as "normal" between 0-7, "mild" at 8-9, "moderate" at 10-12, severe at 13-16 and extremely severe at 17 or more
Change from Week 4 in Depression, Anxiety, Stress Score (DASS-21) and Week 8 | Week 4 and Week 8
  DASS-21 has twenty-one questions, and is a self-administered survey, measuring core symptoms associated with depression, anxiety, and stress on a four-point Likert scale to indicate each symptom's frequency and intensity for the past week. Ratings begin at 0 as "Never" to 3 for "Almost Always". Depression is interpreted as "normal" when the score is between 0-4, mild at 5-6, moderate at 7-10, severe at 11-13 and extremely severe at 14+. Anxiety is categorised as normal between 0-3, mild at 4-5, moderate at 6-7, severe at 8-9 and extremely severe at 10 or more. Stress is indicated as "normal" between 0-7, "mild" at 8-9, "moderate" at 10-12, severe at 13-16 and extremely severe at 17 or more
Change from Week 4 in Depression, Anxiety, Stress Score (DASS-21) and Week 10 | Week 4 and Week 10
  DASS-21 has twenty-one questions, and is a self-administered survey, measuring core symptoms associated with depression, anxiety, and stress on a four-point Likert scale to indicate each symptom's frequency and intensity for the past week. Ratings begin at 0 as "Never" to 3 for "Almost Always". Depression is interpreted as "normal" when the score is between 0-4, mild at 5-6, moderate at 7-10, severe at 11-13 and extremely severe at 14+. Anxiety is categorised as normal between 0-3, mild at 4-5, moderate at 6-7, severe at 8-9 and extremely severe at 10 or more. Stress is indicated as "normal" between 0-7, "mild" at 8-9, "moderate" at 10-12, severe at 13-16 and extremely severe at 17 or more
Change from Week 10 in Depression, Anxiety, Stress Score (DASS-21) at 1-month follow-up | Week 10 and 1-month follow-up
  DASS-21 has twenty-one questions, and is a self-administered survey, measuring core symptoms associated with depression, anxiety, and stress on a four-point Likert scale to indicate each symptom's frequency and intensity for the past week. Ratings begin at 0 as "Never" to 3 for "Almost Always". Depression is interpreted as "normal" when the score is between 0-4, mild at 5-6, moderate at 7-10, severe at 11-13 and extremely severe at 14+. Anxiety is categorised as normal between 0-3, mild at 4-5, moderate at 6-7, severe at 8-9 and extremely severe at 10 or more. Stress is indicated as "normal" between 0-7, "mild" at 8-9, "moderate" at 10-12, severe at 13-16 and extremely severe at 17 or more
Change from 1-month follow-up in Depression, Anxiety, Stress Score (DASS-21) at 3-month follow-up | 1-month follow-up and 3-month follow-up
  DASS-21 has twenty-one questions, and is a self-administered survey, measuring core symptoms associated with depression, anxiety, and stress on a four-point Likert scale to indicate each symptom's frequency and intensity for the past week. Ratings begin at 0 as "Never" to 3 for "Almost Always". Depression is interpreted as "normal" when the score is between 0-4, mild at 5-6, moderate at 7-10, severe at 11-13 and extremely severe at 14+. Anxiety is categorised as normal between 0-3, mild at 4-5, moderate at 6-7, severe at 8-9 and extremely severe at 10 or more. Stress is indicated as "normal" between 0-7, "mild" at 8-9, "moderate" at 10-12, severe at 13-16 and extremely severe at 17 or more

SECONDARY OUTCOMES:
Positive Mental Health (PMH-19) to Week 0 | Week 0
  This 19-item instrument was developed and tested by the IMH research team to assess the six dimensions of positive mental health in Singapore's multi-ethnic population. subscales consist of General Coping (2-items), Emotional support (3-items), Spirituality (4-items), Interpersonal skills (3-items), Personal Growth & Autonomy (4-items), Global affect (3-items). Participants will select on a scale of 1 (not at all like me) to 6 (exactly like me) for the first five subscales. On the 6th subscale, participants indicate how frequently they felt over the past month on a five-point response scale. Scores are added over each subscale and divided by the number of items in that subscale. Higher subscale scores indicate a higher PMH.
Change from Baseline in Positive Mental Health (PMH-19) to Week 4 | Week 0 and Week 4
  This 19-item instrument was developed and tested by the IMH research team to assess the six dimensions of positive mental health in Singapore's multi-ethnic population. subscales consist of General Coping (2-items), Emotional support (3-items), Spirituality (4-items), Interpersonal skills (3-items), Personal Growth & Autonomy (4-items), Global affect (3-items). Participants will select on a scale of 1 (not at all like me) to 6 (exactly like me) for the first five subscales. On the 6th subscale, participants indicate how frequently they felt over the past month on a five-point response scale. Scores are added over each subscale and divided by the number of items in that subscale. Higher subscale scores indicate a higher PMH.
Change from Week 4 in Positive Mental Health (PMH-19) up to Week 8 | Week 4 up to Week 8
  This 19-item instrument was developed and tested by the IMH research team to assess the six dimensions of positive mental health in Singapore's multi-ethnic population. subscales consist of General Coping (2-items), Emotional support (3-items), Spirituality (4-items), Interpersonal skills (3-items), Personal Growth & Autonomy (4-items), Global affect (3-items). Participants will select on a scale of 1 (not at all like me) to 6 (exactly like me) for the first five subscales. On the 6th subscale, participants indicate how frequently they felt over the past month on a five-point response scale. Scores are added over each subscale and divided by the number of items in that subscale. Higher subscale scores indicate a higher PMH.
Change from Week 4 in Positive Mental Health (PMH-19) up to Week 10 | Week 4 up to Week 10
  This 19-item instrument was developed and tested by the IMH research team to assess the six dimensions of positive mental health in Singapore's multi-ethnic population. subscales consist of General Coping (2-items), Emotional support (3-items), Spirituality (4-items), Interpersonal skills (3-items), Personal Growth & Autonomy (4-items), Global affect (3-items). Participants will select on a scale of 1 (not at all like me) to 6 (exactly like me) for the first five subscales. On the 6th subscale, participants indicate how frequently they felt over the past month on a five-point response scale. Scores are added over each subscale and divided by the number of items in that subscale. Higher subscale scores indicate a higher PMH.
Change from Week 10 in Positive Mental Health (PMH-19) at 1-month follow-up | Week 10 and 1-month follow-up
  This 19-item instrument was developed and tested by the IMH research team to assess the six dimensions of positive mental health in Singapore's multi-ethnic population. subscales consist of General Coping (2-items), Emotional support (3-items), Spirituality (4-items), Interpersonal skills (3-items), Personal Growth & Autonomy (4-items), Global affect (3-items). Participants will select on a scale of 1 (not at all like me) to 6 (exactly like me) for the first five subscales. On the 6th subscale, participants indicate how frequently they felt over the past month on a five-point response scale. Scores are added over each subscale and divided by the number of items in that subscale. Higher subscale scores indicate a higher PMH.
Change from 1-month follow-up in Positive Mental Health (PMH-19) at 3-month follow-up | 1-month follow-up and 3-month follow-up
  This 19-item instrument was developed and tested by the IMH research team to assess the six dimensions of positive mental health in Singapore's multi-ethnic population. subscales consist of General Coping (2-items), Emotional support (3-items), Spirituality (4-items), Interpersonal skills (3-items), Personal Growth & Autonomy (4-items), Global affect (3-items). Participants will select on a scale of 1 (not at all like me) to 6 (exactly like me) for the first five subscales. On the 6th subscale, participants indicate how frequently they felt over the past month on a five-point response scale. Scores are added over each subscale and divided by the number of items in that subscale. Higher subscale scores indicate a higher PMH.
Self-Compassion Scale-Short Form (SCS-SF12) to Week 0 | Week 0
  12-item measure, six domains: self-kindness, self-judgment, common humanity, isolation, mindfulness, and over-identification. There are 2-items for each domain. Participants indicate on each item, in response to, "How I typically act towards myself in difficult times", from the 5-point Likert scale ranging from 1 being "almost never" to 5 being "almost always". subscales calculate scores to identify domains to improve. An overall score will also be calculated, with the average score being three and the cut off being five.
  In the domains of self-judgment, isolation, and over-identification, scores higher than 3 indicates lesser self-compassion. In self-kindness, common humanity and mindfulness, scores above 3 indicate higher self-compassion.
Change from Baseline in Self-Compassion Scale-Short Form (SCS-SF12) to Week 4 | Week 0 and Week 4
  12-item measure, six domains: self-kindness, self-judgment, common humanity, isolation, mindfulness, and over-identification. There are 2-items for each domain. Participants indicate on each item, in response to, "How I typically act towards myself in difficult times", from the 5-point Likert scale ranging from 1 being "almost never" to 5 being "almost always". subscales calculate scores to identify domains to improve. An overall score will also be calculated, with the average score being three and the cut off being five.
  In the domains of self-judgment, isolation, and over-identification, scores higher than 3 indicates lesser self-compassion. In self-kindness, common humanity and mindfulness, scores above 3 indicate higher self-compassion.
Change from Week 4 in Self-Compassion Scale-Short Form (SCS-SF12) at Week 10 | Week 4 and Week 10
  12-item measure, six domains: self-kindness, self-judgment, common humanity, isolation, mindfulness, and over-identification. There are 2-items for each domain. Participants indicate on each item, in response to, "How I typically act towards myself in difficult times", from the 5-point Likert scale ranging from 1 being "almost never" to 5 being "almost always". subscales calculate scores to identify domains to improve. An overall score will also be calculated, with the average score being three and the cut off being five.
  In the domains of self-judgment, isolation, and over-identification, scores higher than 3 indicates lesser self-compassion. In self-kindness, common humanity and mindfulness, scores above 3 indicate higher self-compassion.
Change from Week 10 in Self-Compassion Scale-Short Form (SCS-SF12) at 1-month follow-up | Week 10 and 1-month follow-up
  12-item measure, six domains: self-kindness, self-judgment, common humanity, isolation, mindfulness, and over-identification. There are 2-items for each domain. Participants indicate on each item, in response to, "How I typically act towards myself in difficult times", from the 5-point Likert scale ranging from 1 being "almost never" to 5 being "almost always". subscales calculate scores to identify domains to improve. An overall score will also be calculated, with the average score being three and the cut off being five.
  In the domains of self-judgment, isolation, and over-identification, scores higher than 3 indicates lesser self-compassion. In self-kindness, common humanity and mindfulness, scores above 3 indicate higher self-compassion.
Change from 1-month follow-up in Self-Compassion Scale-Short Form (SCS-SF12) at 3-month follow-up | 1-month follow-up and 3-month follow-up
  12-item measure, six domains: self-kindness, self-judgment, common humanity, isolation, mindfulness, and over-identification. There are 2-items for each domain. Participants indicate on each item, in response to, "How I typically act towards myself in difficult times", from the 5-point Likert scale ranging from 1 being "almost never" to 5 being "almost always". subscales calculate scores to identify domains to improve. An overall score will also be calculated, with the average score being three and the cut off being five.
  In the domains of self-judgment, isolation, and over-identification, scores higher than 3 indicates lesser self-compassion. In self-kindness, common humanity and mindfulness, scores above 3 indicate higher self-compassion.
Acceptability of Intervention Measure (AIM) | Week 4
  4-item psychometric measure used to assess perceived acceptability. Participants indicate on the five-point Likert scale from "Completely Disagree" to "Completely Agree". The score is calculated by averaging the response.
Change from Week 4 in Acceptability of Intervention Measure (AIM) Week 10 | Week 4 and Week 10
  4-item psychometric measure used to assess perceived acceptability. Participants indicate on the five-point Likert scale from "Completely Disagree" to "Completely Agree". The score is calculated by averaging the response.
Intervention Appropriateness Measure (IAM) | Week 4
  4-item psychometric measure used to assess perceived appropriateness. Participants indicate on the five-point Likert scale from "Completely Disagree" to "Completely Agree". The score is calculated by averaging the response.
Change from Week 4 in Intervention Appropriateness Measure (IAM) Week 10 | Week 4 and Week 10
  4-item psychometric measure used to assess perceived appropriateness. Participants indicate on the five-point Likert scale from "Completely Disagree" to "Completely Agree". The score is calculated by averaging the response.
Feasibility of Intervention Measure (FIM) | Week 4
  4-item psychometric measure used to assess perceived feasibility of treatment. Participants indicate on the five-point Likert scale from "Completely Disagree" to "Completely Agree". The score is calculated by averaging the response.
Change from Week 4 in Feasibility of Intervention Measure (FIM) and Week 10 | Week 4 and Week 10
  4-item psychometric measure used to assess perceived feasibility of treatment. Participants indicate on the five-point Likert scale from "Completely Disagree" to "Completely Agree". The score is calculated by averaging the response.

OTHER OUTCOMES:
Focus Group Discussions (FGD) | 3-month post-intervention
  Participants' experience will be recorded during the focus group discussion, guided by the semi-structured questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jamilah H Abdul Khaiyom, PhD, Principal Investigator — International Islamic University Malaysia
Locations (2):
- Singapore (2):
  - PERGAS, Singapore
  - Club HEAL, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Grensman A, Acharya BD, Wandell P, Nilsson GH, Falkenberg T, Sundin O, Werner S. Effect of traditional yoga, mindfulness-based cognitive therapy, and cognitive behavioral therapy, on health related quality of life: a randomized controlled trial on patients on sick leave because of burnout. BMC Complement Altern Med. 2018 Mar 6;18(1):80. doi: 10.1186/s12906-018-2141-9. PMID 29510704
- [Result] Zemestani M, Fazeli Nikoo Z. Effectiveness of mindfulness-based cognitive therapy for comorbid depression and anxiety in pregnancy: a randomized controlled trial. Arch Womens Ment Health. 2020 Apr;23(2):207-214. doi: 10.1007/s00737-019-00962-8. Epub 2019 Apr 13. PMID 30982086
- [Result] Chan SHW, Chan WWK, Chao JYW, Chan PKL. A randomized controlled trial on the comparative effectiveness of mindfulness-based cognitive therapy and health qigong-based cognitive therapy among Chinese people with depression and anxiety disorders. BMC Psychiatry. 2020 Dec 14;20(1):590. doi: 10.1186/s12888-020-02994-2. PMID 33317481